CLINICAL TRIAL: NCT06868563
Title: Motor and Sensory Nerve Conduction Studies in Amateur Football, Volleyball and Tennis Athletes
Brief Title: Nerve Conduction Studies in Amateur Football, Volleyball and Tennis Athletes
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Umut Paksoy, Lecturer, Istanbul Bilgi University
Other Study IDs: 2024/09
Record Dates: First submitted 2025-02-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Volleyball Players; Football Players
Keywords: EMG; nerve conduction studies; nerve conduction velocity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control Group: Participants in this group were selected from individuals who had not actively participated in any sports training or competition in the past year.
  Nerve conduction studies were performed on the ulnar sensory, median motor, tibial motor, and sural sensory nerves for both the dominant and non-dominant extremities of the participants using an EMG device.
- Football Group: Participants in this group were selected from athletes who have been actively engaged in sports for the past year and have participated in football training or competitions at least three times a week, for a total of at least 6 hours.
  Nerve conduction studies were performed on the ulnar sensory, median motor, tibial motor, and sural sensory nerves in both the dominant and non-dominant extremities of the participants using an EMG device.
- Volleyball Group: Participants in this group were selected from athletes who have been actively engaged in sports for the past year and have participated in volleyball training or competitions at least three times a week, for a total of at least 6 hours.
  Nerve conduction studies were performed on the ulnar sensory, median motor, tibial motor, and sural sensory nerves in both the dominant and non-dominant extremities of the participants using an EMG device.
- Tennis Group: Participants in this group were selected from athletes who have been actively engaged in sports for the past year and have participated in tennis training or competitions at least three times a week, for a total of at least 6 hours.
  Nerve conduction studies were performed on the ulnar sensory, median motor, tibial motor, and sural sensory nerves in both the dominant and non-dominant extremities of the participants using an EMG device.

SUMMARY:
The aim of the study was to determine how nerve conduction velocities in the upper and lower extremities of athletes in football, volleyball and tennis branches change. The study was completed with a total of 64 participants in 4 groups, with equal numbers of participants in the groups: football, volleyball and tennis players, and a control group that does not do sports. Nerve conduction studies (ulnar sensory, median motor, tibial motor and sural sensory nerves) with an EMG (electromyography) device were applied to participants in 4 groups.

DETAILED DESCRIPTION:
The nerve conduction studies in the research were conducted using a Neuro-MEP-4 branded 4-channel digital EMG/EP (electromyography/evoked potentials) device manufactured by Neurosoft. Throughout the measurements, various equipment was used, including ring electrodes, grounding electrodes, stimulation electrodes, recording electrodes, electrode fixation straps, a marker pen for marking, a measuring tape for distance measurement, ultrasound gel for conductivity, skin disinfectant and paper towels for cleaning, and a pillow for positioning. The measurements were carried out in an electroneurophysiology laboratory that provided a quiet and artifact-free isolated environment.

To facilitate the measurements, participants were requested to wear clothing that could be rolled up to the knee and elbow area. Before the measurements, it was checked whether the participants had been fasting or dehydrated for an extended period. If such a condition was detected, their hunger and dehydration were addressed to prevent nerve conduction changes due to hyponatremia. Additionally, participants were asked to remove accessories such as rings, watches, and bracelets, and electronic devices, including mobile phones, were kept outside the laboratory. If the participants had cold hands or feet, their extremities were warmed using a heater to avoid any impact on nerve conduction. Furthermore, to prevent potential risks, participants were asked whether they had a pacemaker or a history of epilepsy.

Upper extremity nerve measurements were conducted while participants were seated with pillow support, while lower extremity nerve measurements were taken with participants in supine and prone positions on the examination table. The average skin temperature was 32.2°C, ranging between 31-33°C. Participants with cold skin temperatures had their extremities warmed using an infrared heat lamp. The average room temperature was 26.3°C. All participants were tested at the same time of day in the morning to eliminate the effects of circadian rhythm, and they were advised to avoid strenuous physical activity on the test day.

For the median motor nerve conduction study, the participant was positioned on a chair with pillow support under the forearm. The participant's clothing was rolled up above the elbow, and all accessories were removed. The skin area to be measured was cleaned, and gel was applied to the recording electrode, which was then placed on the abductor pollicis brevis (APB) muscle using the belly-tendon technique. The ground electrode was placed between the stimulation and recording electrodes.

The participant was instructed to relax their muscles, and initially, a low-intensity stimulation of 10 milliampere (mA) was applied at the distal stimulation site (approximately 8 centimeter (cm) proximally from the active recording electrode, at the wrist, between the flexor carpi radialis (FCR) and palmaris longus (PL) tendons, and 2 cm proximal to the distal wrist crease) after applying gel to the stimulation electrode. The current intensity was gradually increased to a supramaximal level, and the compound muscle action potential (CMAP) response was recorded. The best response was identified, and the distal stimulation site was marked with a marker pen. The distance between the recording electrode and the distal stimulation site was measured with a measuring tape and recorded.

Next, stimulation was applied at the proximal stimulation site (at the antecubital fossa, just medial to the biceps tendon). The stimulation intensity was increased to a supramaximal level, and the CMAP response was obtained. The proximal stimulation site was also marked with a marker pen. The distance between the proximal and distal stimulation sites was measured with a measuring tape and recorded.

The latency and amplitude values of the recorded CMAP responses were automatically calculated and recorded by the EMG software. The distances measured with the measuring tape were entered into the EMG software, and the nerve conduction velocities were calculated. The measurements were performed on both the right and left extremities.

For the ulnar nerve sensory conduction study, the participant was positioned on a chair with a pillow placed under the forearm for support. The participant's clothing was rolled up to expose the area above the elbow. Accessories were removed, and the skin area to be measured was cleaned. The participant was instructed to keep their extremity relaxed while positioning the forearm in maximal supination with internal rotation of the arm.

The ulnar nerve sensory conduction study was performed using the antidromic method. Ring electrodes were placed on the 5th finger with the black electrode proximally and the red electrode distally after applying gel. The ground electrode was fixed to the palm. The stimulation electrode was positioned 11-13 cm proximally from the active recording electrode, lateral to the flexor carpi ulnaris (FCU) tendon, after applying gel. The conduction study was initiated with a low-intensity current of 2 mA, and the stimulus intensity was gradually increased until an appropriate sensory nerve action potential (SNAP) was obtained. Once a clear SNAP response was observed, stimulation was repeated 5-6 times, and averaging was performed.

Next, the stimulation site was marked with a felt-tip pen, and the distance between the active recording electrode and the stimulation point was measured with a measuring tape and recorded. The latency and amplitude data of the SNAP response obtained from averaging were recorded in the EMG software. After entering the measured distance between the stimulation and recording electrodes into the program, the sensory conduction velocity of the ulnar nerve was determined. All procedures were performed for both the right and left extremities.

For the tibial nerve motor conduction study, the participant was positioned in a supine position on the examination table. The participant was asked to roll up their clothing above the knee level, and accessories were removed. The extremity was cleaned before the procedure.

The recording electrode was placed on the abductor hallucis muscle using the belly-tendon technique with gel and was securely fixed. The ground electrode was placed in an area between the stimulation and recording electrodes. The participant was instructed to keep their muscles relaxed. For distal stimulation, the stimulator electrode was placed approximately 8 cm proximally from the active recording electrode, on the posterior side of the medial malleolus, after applying gel. An initial low-intensity stimulation of 10 mA was applied, then gradually increased to a supramaximal level. The resulting CMAP response was recorded. The distal stimulation point was marked with a felt-tip pen, and the distance between the active recording electrode and the distal stimulation site was measured with a tape measure and recorded.

For proximal stimulation, the participant's knee was positioned at a 30-45° flexion angle, and they were instructed to keep their muscles relaxed. The stimulator electrode was placed on the popliteal fossa with gel. While placing the stimulation electrode, the examiner provided support under the participant's knee to ensure muscle relaxation and obtain a good response. Due to the deep location of the nerve in this region, in muscular participants, both the stimulus intensity and duration were increased to obtain a response. The supramaximal stimulation was applied, and the resulting CMAP response was recorded.

The latency and amplitude values of the CMAP response were automatically generated in the EMG software. The proximal stimulation site was then marked with a felt-tip pen, and the distance between the proximal and distal stimulation sites was measured with a tape measure and recorded. After entering these distance values into the program, the motor conduction velocity of the tibial nerve was determined. The measurements were performed on both extremities.

For the sural nerve sensory conduction study, the participant was positioned in a prone position on the examination table, ensuring that the ankle remained free for testing. The participant was asked to roll up their clothing above the knee level, and accessories were removed. The extremity was cleaned before the procedure.

This study was performed using the antidromic method. The recording electrode was placed behind the lateral malleolus after applying gel. The ground electrode was positioned and secured between the stimulation and recording electrodes. The stimulation electrode was placed approximately 12-14 cm proximally from the active recording electrode, lateral to the midline of the calf, after applying gel.

The participant was instructed to keep their muscles relaxed, and a low-intensity stimulation of 2 mA was applied. The stimulus intensity was gradually increased until an appropriate SNAP response was obtained. Once a clear SNAP response was recorded, 5-6 additional stimulations were applied, and averaging was performed.

The latency and amplitude values of the SNAP response obtained from averaging were recorded in the EMG software. The stimulation site was then marked with a felt-tip pen, and the distance between the active recording electrode and the stimulation site was measured with a tape measure and recorded. After entering the measured distances into the program, the nerve conduction velocity of the sural nerve was determined. All procedures were performed for both extremities.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old and under 35 years old,
* Being willing to participate in the study,
* Signing the informed consent form,
* Athlete groups must have been actively training for at least 3 days per week and a minimum of 6 hours per week over the past year,

Exclusion Criteria:

* Being under 18 and over 35
* Having metabolic diseases that may affect nerve conduction speeds (hypothyroidism, hyperthyroidism, diabetes mellitus, etc.)
* Participants who are not suitable for EMG measurement, such as cardiac problems, skin infections, and epilepsy
* Having had a previous surgical operation on the extremity where EMG measurement will be performed

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy adult individuals divided into four groups: sedentary individuals (control group), football players, volleyball players, and tennis players. Participants were recruited from local sports clubs, university teams, and recreational athletes. The control group consists of individuals who have not engaged in regular sports activities. All participants were assessed in a single session at a designated laboratory setting.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Electromyography | One-time assessment on the day of enrollment, approximately 1 hour per participant.
  It was performed with a 4-channel digital EMG/EP device, branded as Neuro-MEP-4, a Neurosoft company. Equipment such as ring electrode, grounding electrode, stimulation electrode, recording electrode, electrode fixation velcro, felt-tip pen for marking, tape measure for distance measurement, ultrasound gel for providing conductivity, skin disinfectant and paper towel for cleaning, and pillow for positioning were used throughout the measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Bilgi University Electroneurophysiology Laboratory, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No